CLINICAL TRIAL: NCT03235596
Title: Pilot Study Investigating the Effects of Cathodal Transcranial Direct Current Stimulation (tDCS) on Executive Functions of Patients With Autism Without Mental Retardation. TRANSFEX Study
Brief Title: Effects of Cathodal tDCS on Executive Functions in Autism
Acronym: TRANSFEX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier du Rouvray (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-A00805-46
Record Dates: First submitted 2017-06-21; First posted 2017-08-01 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-06

CONDITIONS: Autism Spectrum Disorder
Keywords: executive functions; tDCS
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: It's an interventional, prospective and monocentric pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treated arm (Experimental): Patients received cathodal tDCS applied over the left dorsolateral prefrontal cortex at 2 mA during 15 minutes. They have 10 sessions in 5 consecutive days, 2 sessions per day.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — cathodal tDCS applied over the left dorsolateral prefrontal cortex at 2mA during 15 minutes

SUMMARY:
It's an interventional, prospective and monocentric pilot study concerning adult patients with autism without mental retardation.

The primary outcome is to assess the effects of cathodal transcranial direct current stimulation (tDCS) on the left dorsolateral prefrontal cortex (DLPFC) on the executive functions of patients with autism without mental retardation or with Asperger syndrome.

The secondary outcomes are to evaluate the safety of this treatment and to evaluate its impact on impaired social communication and on restricted or repetitive behaviors.

DETAILED DESCRIPTION:
The patients concerned by the study are aged 20 to 50 years old. They meet ICD-10 criteria for autism without mental retardation or Asperger syndrome and they have adaptive capacity and autonomy complaints. They stable treatments for at least 4 weeks prior and during all the study and no history of tDCS. Women of childbearing age with no adequate contraception, pregnant or lactating women are excluded.

This is an interventional, prospective and monocentric pilot study. The patient is informed about the clinical study during the psychiatric consultation. The patient is provided with a cooling-off period of several days. During the inclusion visit, the executive functions of the patient are assessed (WSCT, Stroop, TMT A and B and verbal fluency test). If 2 pathological tests are found among all measured scores: administration of ISDC and EC2R (interview of the person accompanying) and planning of the first tDCS session 15 days later. If no pathological test is found : study exit.

The treatment consists in 10 sessions of cathodal tDCS applied over the left dorsolateral prefrontal cortex (DLPFC) at 2mA. Each session lasts 15 minutes. They are 2 sessions per day.

Ten days after the end of tDCS treatment, patients are assessed for executive functions and behavioral dysexecutive functions (EC2R and ISCD).

ELIGIBILITY:
Inclusion Criteria:

* With ICD-10 criteria for autism without mental retardation or Asperger syndrome;
* Patient with adaptive capacity and autonomy complaints.
* Patients with stable treatments for at least 4 weeks prior and during all the study;
* Patient with no history of tDCS;
* Patients affiliated to a social security system;
* Patients who give their informed written consents;
* For women of childbearing age: effective contraception; required (estrogen and progestogen or intra-uterine device or tubal ligation) for at least 1 month before starting treatment (a negative pregnancy test has been obtained).

Exclusion Criteria:

* Skin disease, dementia, history of epileptic seizures, brain tumor or metallic implants/implanted electrical devices.
* Patients who followed à cognitive remediation program during the last 6 months;
* Subjects currently treated with magnetic or electrical stimulation techniques (e.g.: transcutaneous or root stimulation).
* Women of childbearing age with no adequate contraception, pregnant or lactating women;
* Patients participating or having participated in an interventional clinical trial within 30 days prior to the inclusion visit;
* Subjects who are deprived of their liberty by decision of a judicial or administrative authority.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Cognitive dysexecutive functions | 30 days
  Score changes in Wisconsin Card Sorting test between assessment at day 1(inclusion) and assessment at day 30 (end of the study).

SECONDARY OUTCOMES:
Score changes in the tDCS adapted version of the Udvalg pour Kliniske Undersøgelser (UKU) Side Effect Rating Scale | 30 days
  Score changes in the tDCS adapted version of the Udvalg pour Kliniske Undersøgelser (UKU) Side Effect Rating Scale between assessment at day 1 (inclusion), assessment at day 20 and assessment day 30 (end of the study).
Behavioral dysexecutive functions | 30 days
  Score changes in the behavioral dysexecutive syndrome battery (Inventaire du Syndrome Dysexécutif Comportemental, ISDC) and the restricted and repetitive behaviors rating scale (Echelle d'évaluation des Comportements Répétitifs et Restreints, EC2R) between assessment at day 1 (inclusion) and assessment at day 30 (end of the study) (interview of the person accompanying).
Trail Making Test A and B | 30 days
  Score changes in the Trail Making test A and B between assessment at day 1 (inclusion) and assessment at day 30 (end of the study).
Stroop Test | 30 days
  Score changes in the Stroop between assessment at day 1 (inclusion) and assessment at day 30 (end of the study).
Verbal Fluency Test | 30 days
  Score changes in Verbal Fluency Test between assessment at day 1 (inclusion) and assessment at day 30 (end of the study).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier du Rouvray, Sotteville-lès-Rouen, France

IPD SHARING:
Plan to Share IPD: No